CLINICAL TRIAL: NCT06125873
Title: Effect of Moringa Leaf Capsules on Glycemic Control of Type 2 Diabetic Patients- an Interventional Study
Brief Title: Effect of Moringa Leaf Capsules on Glycemic Control of Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Islamabad Medical and Dental College (Other)
Responsible Party: Principal Investigator, Professor Dr. Asma Irfan, Professor and Head of Department, Islamabad Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: imdc123; No 99/IMDDC/IRB-2022 (Other Grant/Funding Number: IMDC)
Record Dates: First submitted 2023-03-29; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2; Moringa Leaf powder; Side effects
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Metformin 500mg taken orally twice daily
  Interventions: Drug: Metformin
- "Moringa+Metformin" (Experimental): Metformin 500mg taken orally twice daily with Moringa Oliefera (MO) capsule 1g once daily before breakfast
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Moringa + Metformin - Moringa 1 gm and Metformin 500 mg
  Other Names: Metformin is a glucose-lowering drug by inhibiting hepatic gluconeogenesis and opposing the action of glucagon.

SUMMARY:
A randomized clinical trial will be done on 50 patients , randomly divided into two groups by lottery method to compare the glycemic control in patients of Type 2 Diabetes Mellitus by the use of Moringa Oleifera (MO) capsules. Patients will be given Moringa Oleifera (MO) capsules for 3 months and follow up will be conducted after 3 months to assess glycemic control.

DETAILED DESCRIPTION:
Few human studies are reported on Moringa Oleifera (MO), with most trials reported on animals. Based on human studies, the plant has been proposed to decrease glucose levels by increasing insulin secretion and sensitivity and by inhibiting amylase and glucosidase activities proven by animal studies, additional proposed mechanisms of action include increased glucose uptake in the muscle and liver, inhibition of glucose uptake in the intestine, and decreased gluconeogenesis in the liver.

Rationale of this study is to observe the effects of Moringa Oleifera (MO) capsules, a herbal medicine, on lowering Hba1c levels and compare it with the first line drug so that it can be recommended in the guidelines as a supportive treatment option.

A few human studies are reported on the use of Moringa Oleifera (MO), most of trials are reported on animals. In Pakistan no such study is available but people in rural areas take it as a myth to treat different diseases.

Moringa Oleifera (MO) leaves are non-toxic. This has been confirmed by laboratory experiments such as The aqueous extract of leaves was administered orally to 30 male Wistar rats and even in doses of 2000 mg/kg no mortality ensued. Sub-acute toxicity was assessed by administering daily doses of up to 1600 mg kg to male rats, and no signs of serious toxicity were observed on biochemical or haematological tests, or on histopathology of the organs.

According to the International Diabetes Federation, in the year 2022, 26.7% of adults in Pakistan are a victim of diabetes mellitus, making the total number of cases approximately 33,000,000. This alarmingly high number poses not only an enormous risk of health complications but also a huge financial load on patients. A substantial proportion of patients' income is spent on diabetes care. The mean annual direct cost per patient with diabetes was estimated to be 80,000 Rupees. Medications accounted for the largest share (60.4%) of this cost. The WHO has supported the evaluation of medicinal plants and herbs for the management of certain chronic conditions. In recent years there has been exponential growth in the field of herbal medicines and the demand for these is increasing both in developing and developed countries because of their natural origin, fewer side effects and low cost.

The objective of this study is to assess the combined effect of metformin and Moringa Oleifera (MO) capsules on the participants of glycaemic control (Type 2 diabetics), the safety of Moringa Oleifera (MO) capsules by measuring the partcipant's Liver function tests(LFTs) and Renal function tests(RFTs). HbA1c level of ≥ 7.0% will be considered as 'poor glycemic control'.

Pilot testing will be done on 5% of the sample before conducting the whole study.Informed written consent will be taken from the enrolled patients and confidentiality will be maintained throughout the study. A detailed history will be taken focusing on duration and onset, family history, lifestyle and daily activities. Liver Function Tests and Renal Function Tests will be assessed. A questionnaire attached will be used by the investigators for taking participant's history, anthropometric measures, and demographic details. Data will be collected under the supervision of a diabetic specialist. Particpants will be requested to visit ANTH hospital every month to get their lab investigations done and to report side effects if any. Glycated haemoglobin (HbA1c) will be determined by high-performance liquid chromatography before and at the end of the study by a skilled Lab technician in (ANTH). Fasting blood glucose levels will be measured by a glucometer and participants will also be instructed and guided on the first visit to use a glucometer to check and note daily fasting glucose levels. The questions regarding any side effects are included in the questionnaire. There will be no potential risk to the patient, as monitoring of RFTs, LFTs, and Lipid profiles will be done every month. If lab reports are deranged on participant's first visit to the hospital, participant will be excluded from the study. Random distribution of patients will be done through lottery method. Group A will be treated with Tablet Metformin 500mg twice a day and group B with Moringa Oleifera (MO) capsules along with patients usual dose of Tablet Metformin. All the patients will be advised to have proper diet control and lifestyle modifications.

The data will be analyzed with the help of Statistical Package for Social Sciences (SPSS) version 25. Chi-square test will be applied to compare the clinical efficacy, and safety in terms of any side effect between both groups throughout the study period. P-value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:• The patients of over age 40 with type 2 diabetes

* The patients who willingly consent

Exclusion Criteria:• Patients having Type I diabetes

* Pregnant women
* The patients with deranged LFTs and RFTs.
* Patients having Creatinine levels more than 1.3 mg/dl in man and >1.1mg/dl in female.
* Patients of Type II diabetes on insulin therapy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Moringa leaf powder decreases blood sugar level in type 2 diabetic patients. | 3 months
  Fasting blood glucose tested after 15 days regularly.
It controls blood Glycated hemoglobin level in type 2 diabetic patients. | 3 months
  Glycated Hemoglobin(Hb A1c) tested after 3 months.

SECONDARY OUTCOMES:
Moringa leaf powder effect on Systolic Blood Pressure | 3 months
  Systolic BP will be measured in mm Hg at the start of study and then after every 3 months
Moringa leaf powder effect on Diastolic Blood Pressure | 3 months
  Diastolic BP will be measured in mm Hg at the start of study and then after every 3 months
Moringa leaf powder effect on body weight of patients | 3 months
  The weight in kg at the start of study and then after every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yasiri Niazi, MD, Study Director — IMDC
Locations (1):
- Islamabad Medical and Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Result] Azeem S, Khan U, Liaquat A. The increasing rate of diabetes in Pakistan: A silent killer. Ann Med Surg (Lond). 2022 Jun 3;79:103901. doi: 10.1016/j.amsu.2022.103901. eCollection 2022 Jul. No abstract available. PMID 35860160
- [Result] Gillani AH, Aziz MM, Masood I, Saqib A, Yang C, Chang J, Mohamed Ibrahim MI, Fang Y. Direct and indirect cost of diabetes care among patients with type 2 diabetes in private clinics: a multicenter study in Punjab, Pakistan. Expert Rev Pharmacoecon Outcomes Res. 2018 Dec;18(6):647-653. doi: 10.1080/14737167.2018.1503953. Epub 2018 Aug 1. PMID 30052085
- [Result] Owens FS 3rd, Dada O, Cyrus JW, Adedoyin OO, Adunlin G. The effects of Moringa oleifera on blood glucose levels: A scoping review of the literature. Complement Ther Med. 2020 May;50:102362. doi: 10.1016/j.ctim.2020.102362. Epub 2020 Feb 28. PMID 32444043
- [Result] Haber SL, McMahon RP, Barajas J, Hayes AR, Hussein H. Effects of Moringa oleifera in patients with type 2 diabetes. Am J Health Syst Pharm. 2020 Oct 30;77(22):1834-1837. doi: 10.1093/ajhp/zxaa255. No abstract available. PMID 32960218
- [Result] Anthanont P, Lumlerdkij N, Akarasereenont P, Vannasaeng S, Sriwijitkamol A. Moringa Oleifera Leaf Increases Insulin Secretion after Single Dose Administration: A Preliminary Study in Healthy Subjects. J Med Assoc Thai. 2016 Mar;99(3):308-13. PMID 27276742
- [Result] Omar SM, Musa IR, Osman OE, Adam I. Assessment of glycemic control in type 2 diabetes in the Eastern Sudan. BMC Res Notes. 2018 Jun 8;11(1):373. doi: 10.1186/s13104-018-3480-9. PMID 29884216
- [Result] Shahbaz H, Rout P, Gupta M. Creatinine Clearance. 2024 Jul 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK544228/ PMID 31334948
- See also: Type2 diabetes and moringa — https://clinicaltrials.gov

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT06125873/Prot_SAP_ICF_000.pdf